CLINICAL TRIAL: NCT07382050
Title: A Prospective Multicenter Clinical Study on the Efficacy and Safety of the Zirconia Ceramic Hip Joint Prosthesis System After Its Market launchM20251018
Brief Title: A Prospective Multicenter Clinical Study on the Efficacy and Safety of the Zirconia Ceramic Hip Joint Prosthesis System After Its Market Launch
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: Peking Union Medical College Hospital (Other); Peking University First Hospital (Other); Beijing Friendship Hospital (Other); China-Japan Friendship Hospital (Other); Peking University Shougang Hospital (Other); Peking University People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M20251018
Record Dates: First submitted 2026-01-12; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-12

CONDITIONS: THA; Prosthesis
Keywords: total hip arthroplasty; Zirconia ceramic prosthesis; efficacy; safety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Received the hip joint prosthesis system implanted by Beijing Anthrone Technology Co., Ltd.

SUMMARY:
This study adopted a prospective, multi-center, single-group target value trial design to evaluate the safety and efficacy of the hip joint prosthesis system produced by Beijing Anshou Technology Co., Ltd. in total hip arthroplasty. This clinical study selected seven clinical centers and recruited 290 subjects. Each center competed for enrollment, with the requirement that each center should undertake no less than 8 cases and no more than half of the total cases. The enrollment stopped when the total number of cases met the design requirements. After the patients signed the informed consent form, they entered the screening process. After the screening was successful, the hip joint prosthesis system produced by Beijing Anshou Technology Co., Ltd. was implanted, and follow-up was conducted for the patients at "before surgery, on the day of surgery, immediately after surgery until discharge, 2 weeks after surgery, 6 weeks after surgery, 3 months after surgery, 6 months after surgery, and 12 months after surgery." The demographic information and various evaluation indicators of the subjects were collected.

DETAILED DESCRIPTION:
This study adopted a prospective, multi-center, single-group target value trial design to evaluate the safety and efficacy of the hip joint prosthesis system produced by Beijing Anshou Technology Co., Ltd. in total hip arthroplasty. This clinical study selected seven clinical centers and recruited 290 subjects. Each center competed for enrollment, with the requirement that each center should undertake no less than 8 cases and no more than half of the total cases. The enrollment stopped when the total number of cases met the design requirements. After the patients signed the informed consent form, they entered the screening process. After the screening was successful, the hip joint prosthesis system produced by Beijing Anshou Technology Co., Ltd. was implanted, and follow-up was conducted for the patients at "before surgery, on the day of surgery, immediately after surgery until discharge, 2 weeks after surgery, 6 weeks after surgery, 3 months after surgery, 6 months after surgery, and 12 months after surgery." The demographic information and various evaluation indicators of the subjects were collected.

ELIGIBILITY:
Inclusion Criteria:

1. The patient's age ranges from 18 to 80 years old (inclusive), with no gender restrictions.
2. The patient's bones have matured.
3. The patient is indicated for hip replacement surgery
4. The subjects participating in the study were undergoing hip replacement for the first time
5. The subject or his/her guardian is willing and able to sign the informed consent form

Exclusion Criteria:

1. There are contraindications for hip replacement surgery
2. It is known that the patient has a history of allergy to one or more implant materials
3. Pregnant or lactating women
4. Hip dysplasia is classified into CROWE grades 3 and 4
5. Those who are physically weak or unable to tolerate surgery due to other systemic diseases, as well as those with an expected lifespan of less than two years
6. The reasons why other researchers believe that patients are not suitable for this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. The patient's age ranges from 18 to 80 years old (inclusive), with no gender restrictions.
  2. The patient's bones have matured.
  3. The patient is indicated for hip replacement surgery
  4. The subjects participating in the study were undergoing hip replacement for the first time
  5. The subject or his/her guardian is willing and able to sign the informed consent form
Sampling Method: Non-Probability Sample
Enrollment: 290 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Harris score | Six months
  The patient returned to the outpatient department for a follow-up visit, and the scale was followed up

SECONDARY OUTCOMES:
FJS score | Six months
  The patient returned to the outpatient department for a follow-up visit, and the scale was followed up
operation time | Perioperative/Periprocedural
  Measure the time from the moment the knife touches the skin to the completion of the surgical incision suture
WOMAC | Six months
  he patient returned to the outpatient department for a follow-up visit, and the scale was followed up
AE/SAE and postoperative complications | through study completion, an average of 1 year
  Describe the number and frequency of various adverse events, adverse events related to the study product, adverse events leading to dropout, and serious adverse events. Describe the number and frequency of various complications and complications related to the study product. Provide corresponding lists for adverse events and complications. Calculate the survival rate of the prosthesis.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The data will be published in the form of an academic paper.